CLINICAL TRIAL: NCT02284399
Title: National Prevalence and Impact of Noninvasive Prenatal Testing
Status: Completed | Type: Observational
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: OBX0032
Record Dates: First submitted 2014-10-21; First posted 2014-11-06 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Aneuploidy
Keywords: aneuploidy; Trisomy 21; NIPT
MeSH Terms: conditions — Aneuploidy; Down Syndrome | interventions — dichlorobis(azomycin)platinum II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IDTFK Group Post NIPT - (January 2012-June 2014): Pregnant women who present to participating centers between January 2012-June 2014, after the release of non-invasive prenatal testing (NIPT), who are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).
  Interventions: Other: non-invasive prenatal testing
- IDTFK Group pre-NIPT (January 2010-July 2010): A control group of pregnant women, prior to the release of non-invasive prenatal testing (NIPT), who present to participating centers between January 2010-June 2010 and are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).

INTERVENTIONS:
Other: non-invasive prenatal testing — Noninvasive Prenatal Testing (NIPT) of fetal cell free DNA in maternal circulation
  Other Names: NIPT
  Groups: IDTFK Group Post NIPT - (January 2012-June 2014)

SUMMARY:
Information on pregnant women undergoing non-invasive prenatal testing (NIPT) at one of the Obstetrix Medical Groups Outpatient Centers between January 2012 and June 2014 will be retrospectively gathered and an analysis of the impact and prevalence of NIPT. This will be compared to a control group of pregnant women in those same practices undergoing prenatal testing during the months of January 2010-July 2010.

DETAILED DESCRIPTION:
Information regarding the frequency of non-invasive testing (NIPT), the impact of screening on the need for and frequency of invasive testing, and the indications for testing are important for the clinicians in this country to not only understand the impact that this testing has had but also to plan for allocation of personnel and resources in their prenatal testing units, as well as many other more subtle changes including describing changes to referring clinicians and patients and projecting financial impacts. Information on pregnant women undergoing NIPT at one of the Obstetrix Medical Groups Outpatient Centers between January 2012 and June 2014 will be retrospectively gathered and compared to a control group of pregnant women in those same practices undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK) during the months of January 2010-July 2010. An analysis of the impact of NIPT will be done.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* Presented to a participating Obstetrix Outpatient Center for an invasive prenatal diagnostic testing for fetal karyotype (IDTFK) (i.e. amniocentesis or CVS).
* Invasive prenatal diagnostic testing for fetal karyotype (IDTFK) (i.e. amniocentesis or CVS) performed between January 2012 and June 2014 (A control group enrolled between January 2010 - July 2010)

Exclusion Criteria:

* Patient less than 18 years of age
* Patients not receiving a invasive prenatal diagnostic testing for fetal karyotype (IDTFK)(i.e. amniocentesis or CVS) at a participating study center
* Testing NOT done within the window for inclusion (Jan 2012 - June 2014) or Control Group window (January 2010 - July 2010)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women at participating Obstetrix Outpatient centers who are undergoing IDTFK between January 2012 and June 2014.
Sampling Method: Non-Probability Sample
Enrollment: 4488 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06-28 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Maurel, MSN, Study Director — Mednax Inc.
Locations (7):
- United States (7):
  - Phoenix Perinatal Associates, Phoenix, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Maryland Perinatal Associates, Rockville, Maryland
  - Mercy Hospital of St. Louis, St Louis, Missouri
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IDTFK Group Pre-NIPT (January 2010-July 2010): A control group of pregnant women, prior to the release of non-invasive prenatal testing (NIPT), who present to participating centers between January 2010-June 2010 and are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).
  * non-invasive prenatal testing: Noninvasive Prenatal Testing (NIPT) of fetal cell free DNA in maternal circulation.
  * Invasive Diagnostic testing for Fetal Karyotype (IDTFK) = Amniocentesis or chorionic villus sampling (CVS)
- IDTFK Group Post NIPT - (January 2012-June 2014): Pregnant women who present to participating centers between January 2012-June 2014, after the release of non-invasive prenatal testing (NIPT), who are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).
  * non-invasive prenatal testing: Noninvasive Prenatal Testing (NIPT) of fetal cell free DNA in maternal circulation.
  * Invasive Diagnostic testing for Fetal Karyotype (IDTFK) = Amniocentesis or CVS
Period: Overall Study
Arm/Group | IDTFK Group Pre-NIPT (January 2010-July 2010) | IDTFK Group Post NIPT - (January 2012-June 2014)
Started | 1414 | 3074
Completed | 1414 | 3074
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDTFK Group Post NIPT - (January 2012-June 2014) | IDTFK Group Pre-NIPT (January 2010-July 2010) | Total
Number analyzed (Participants) | 3074 | 1414 | 4488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3074 | 1414 | 4488
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3074 | 1414 | 4488
  Male | 0 | 0 | 0
Indication for invasive test was Advance Maternal Age (AMA) [Count of Participants; unit: Participants] | 2071 | 996 | 3067
Indication for invasive test was Family History of Aneuploidy [Count of Participants; unit: Participants] | 304 | 127 | 431
Indication for invasive test was a Positive Serum Screening Test [Count of Participants; unit: Participants] | 995 | 499 | 1494
Indication for invasive test was Ultrasound Abnormality noted [Count of Participants; unit: Participants] | 961 | 292 | 1253
Indication for and invasive test was a Positive cell free DNA (cfDNA) [Count of Participants; unit: Participants] | 133 | 0 | 133
Karyotype Results of Amniocentesis and CVS - Normal Result [Number; unit: indications] — Note: percentages sum to more than 100% because some patient had more than one indication. Population: Note: percentages sum to more than 100% because some patient had more than one indication.
  indications
    Normal karyotype | 2687 | 1310 | 3997
    T21 | 205 | 60 | 265
    T18 | 72 | 19 | 91
    T13 | 24 | 5 | 29
    45X | 34 | 6 | 40
    47XXY | 6 | 4 | 10
    OTHER | 40 | 10 | 50
Indication for an invasive test was multifetal gestation [Count of Participants; unit: Participants] | 76 | 29 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient Undergoing IDTFK Before (Control) and After (Test) NIPT Testing Came to Market
Description: Total Number of patient undergoing invasive diagnostic testing for fetal karyotype (IDTFK) before (control group = Jan - July 2010) and after (test group=Jan 2012-June 2014) NIPT testing came to market
Time Frame: 4 years
Population: This was an observational study that looked to compare the number of patient who underwent IDTFK during Jan 2010-July 2010 (prior to the adoption of NIPT) with the number of patients who underwent IDTFK during Jan 2012-June 2014 (after the adoption of NIPT).
Measure: Count of Participants; unit: Participants
Arm/Group | IDTFK Group Pre-NIPT (January 2010-July 2010) | IDTFK Group Post NIPT - (January 2012-June 2014)
Number analyzed (Participants) | 1414 | 3074
Participants | 1414 | 3074

2. Secondary Outcome: Frequency of Positive Tests for Abnormal Karyotype Before and After the Adoption of NIPT Testing.
Description: Will determine if frequency of positive tests for abnormal karyotypes between the control period and the study period where different.
Time Frame: 4 years
Population: The number of positive tests identified between the control and the test periods.
Measure: Count of Participants; unit: Participants
Groups:
- IDTFK Group Post NIPT - (January 2012-June 2014): Number of pregnant women who present to participating centers between January 2012-June 2014, after the release of non-invasive prenatal testing (NIPT), who are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).
  non-invasive prenatal testing procedure: Noninvasive Prenatal Testing (NIPT) of fetal cell free DNA in maternal circulation
Arm/Group | IDTFK Group Post NIPT - (January 2012-June 2014) | IDTFK Group Pre-NIPT (January 2010-July 2010)
Number analyzed (Participants) | 3074 | 1414
Participants | 454 | 104

ADVERSE EVENTS:
Time Frame: This was an retrospective study. Adverse events were not captured
Description: This was an retrospective study. Adverse events were not captured
Groups:
- IDTFK Group Pre-NIPT (January 2010-July 2010): A control group of pregnant women, prior to the release of non-invasive prenatal testing (NIPT), who present to participating centers between January 2010-June 2010 and are undergoing invasive prenatal diagnostic testing for fetal karyotype (IDTFK).
  * non-invasive prenatal testing: Noninvasive Prenatal Testing (NIPT) of fetal cell free DNA in maternal circulation.
  * Invasive Diagnostic testing for Fetal Karyotype (IDTFK) = Amniocentesis or CVS
Arm/Group | IDTFK Group Pre-NIPT (January 2010-July 2010) | IDTFK Group Post NIPT - (January 2012-June 2014)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes